CLINICAL TRIAL: NCT00883779
Title: A Randomized, Placebo-controlled, Double-blind Phase III Study of the Effect of First-line Treatment With Intercalated Tarceva Versus Placebo in Combination With Gemcitabine/Platinum on Progression-free Survival in Patients With Stage IIIB/IV Non-small Cell Lung Cancer
Brief Title: A Study of Tarceva (Erlotinib) or Placebo in Combination With Platinum-Based Therapy as First Line Treatment in Patients With Advanced or Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MO22201
Record Dates: First submitted 2009-04-15; First posted 2009-04-20 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Cisplatin; Carboplatin; Erlotinib Hydrochloride; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Platinum chemotherapy (cisplatin or carboplatin); Drug: erlotinib [Tarceva]; Drug: gemcitabine
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Platinum chemotherapy (cisplatin or carboplatin); Drug: gemcitabine

INTERVENTIONS:
Drug: Placebo — po on days 15-28 of each 4 week cycle until disease progression
  Arms: 2
Drug: Platinum chemotherapy (cisplatin or carboplatin) — cisplatin --75mg/m2 oon day 1 of each 4 week cycle for 6 cycles or carboplatin--5xAUC on day 1 of each 4 week cycle for 6 cycles
Drug: erlotinib [Tarceva] — 150mg po on days 15-28 of each 4 week cycle until disease progression
  Arms: 1
Drug: gemcitabine — 1250mg/m2 iv on days 1 and 8 of each 4 week cycle for 6 cycles

SUMMARY:
This 2 arm study will compare the efficacy and safety of sequential treatment with Tarceva or placebo, plus platinum-based therapy, as first line treatment in patients with advanced or recurrent non-small cell lung cancer. Patients will be randomized to receive gemcitabine (1250mg/m2 iv) on days 1 and 8, and cisplatin (75mg/m2) or carboplatin (5xAUC)on day 1, followed by Tarceva 150mg/day or placebo from day 15 to day 28 of each 4 week cycle for a total of 6 cycles,then followed by Tarceva or placebo monotherapy.The anticipated time on study treatment is until disease progression, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* advanced (stage IIIB/IV)non-small cell lung cancer;
* measurable disease;
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.

Exclusion Criteria:

* prior exposure to agents directed at the HER axis;
* prior chemotherapy or systemic anti-tumor therapy after advanced disease;
* unstable systemic disease;
* any other malignancy within last 5 years, except cured basal cell cancer of skin or cured cancer in situ of cervix;
* brain metastasis or spinal cord compression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2009-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- China (5):
  - Beijing
  - Guangzhou
  - Hangzhou
  - Nanjing
  - Shanghai
- Hong Kong (2):
  - Hong Kong
  - Shatin
- Indonesia (3):
  - Jakarta
  - Surabaya
  - Yogyakarta
- Philippines (3):
  - Manila
  - Pasig
  - Quezon City
- Gyeonggi-do, South Korea
- Taiwan (2):
  - Taichung
  - Taipei
- Thailand (2):
  - Bangkok
  - Chiang Mai

REFERENCES:
- [Derived] Wu YL, Lee JS, Thongprasert S, Yu CJ, Zhang L, Ladrera G, Srimuninnimit V, Sriuranpong V, Sandoval-Tan J, Zhu Y, Liao M, Zhou C, Pan H, Lee V, Chen YM, Sun Y, Margono B, Fuerte F, Chang GC, Seetalarom K, Wang J, Cheng A, Syahruddin E, Qian X, Ho J, Kurnianda J, Liu HE, Jin K, Truman M, Bara I, Mok T. Intercalated combination of chemotherapy and erlotinib for patients with advanced stage non-small-cell lung cancer (FASTACT-2): a randomised, double-blind trial. Lancet Oncol. 2013 Jul;14(8):777-86. doi: 10.1016/S1470-2045(13)70254-7. Epub 2013 Jun 17. PMID 23782814

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received 1250 milligrams per squared meter (mg/m^2) of gemcitabine intravenous (IV) infusion on Day 1 and 8, carboplatin 5 times (5x) area under concentration versus time curve (AUC) or cisplatin 75 mg/m^2 IV infusion on Day 1 and oral placebo daily from Day 15 to 28 every 4 weeks, continued for 6 cycles (28-day Cycle) until disease progression (PD), unacceptable toxicity or death in primary study treatment phase. Participants who completed 6 cycles of treatment without PD or unacceptable toxicity, or if they withdrew early because of toxicity from platinum-doublet chemotherapy, entered the post-study treatment phase and continued same treatment until PD, unacceptable toxicity or death. Participants who withdrew due to PD or toxicity from placebo could not enter the post-study treatment phase. Upon PD (during either primary or post-study treatment phase), participants had the option to be crossed over to open-label erlotinib 150 mg/day outside the study (Off-study phase).
- Erlotinib: Participants received 1250 mg/m^2 of gemcitabine IV infusion on Day 1 and 8, carboplatin 5x AUC or cisplatin 75 mg/m^2 IV infusion on Day 1 and oral erlotinib 150 milligrams per day (mg/day) from Day 15 to 28 every 4 weeks, continued for 6 cycles (28-day cycle) until PD, unacceptable toxicity or death in the primary study treatment phase. Participants who completed 6 cycles of treatment without PD or unacceptable toxicity, or if they withdrew early because of toxicity from the platinum-doublet chemotherapy, entered the post-study treatment phase and continued same treatment until PD, unacceptable toxicity or death. Participants who withdrew due to PD or toxicity from erlotinib could not enter the post-study treatment phase. Upon PD (during either the primary or post-study treatment phase), participants were treated at the discretion of the investigators' discretion (Off-study phase).
Period: Primary Study Treatment Phase
Arm/Group | Placebo | Erlotinib
Started | 225 | 226
Completed | 120 | 140
Not Completed | 105 | 86
Not completed — Did not receive allocated intervention | 4 | 4
Not completed — Disease progression | 75 | 59
Not completed — Adverse Event | 16 | 16
Not completed — Death | 2 | 3
Not completed — Refused Treatment | 5 | 4
Not completed — Other | 3 | 0
Period: Post-Study Treatment Phase
Arm/Group | Placebo | Erlotinib
Started | 112 | 135
Completed | 0 | 0
Not Completed | 112 | 135
Not completed — Adverse Event | 2 | 3
Not completed — Death | 1 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Refused Treatment | 3 | 0
Not completed — Disease progression | 103 | 122
Not completed — Other | 3 | 0
Not completed — Ongoing in the study | 0 | 6
Period: Off-study Phase
Arm/Group | Placebo | Erlotinib
Started | 209 | 202
Completed | 0 | 0
Not Completed | 209 | 202
Not completed — Death | 185 | 174
Not completed — Refused treatment | 1 | 1
Not completed — Failure to return | 5 | 6
Not completed — Other | 18 | 21

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) population (Included all enrolled participants).
Groups:
- Placebo: Participants received 1250 mg/m^2 of gemcitabine IV infusion on Day 1 and 8, carboplatin 5x AUC or cisplatin 75 mg/m^2 IV infusion on Day 1 and oral placebo daily from Day 15 to 28 every 4 weeks, continued for 6 cycles (28-day cycle) until PD, unacceptable toxicity or death in the primary study treatment phase. Participants who completed 6 cycles of treatment without PD or unacceptable toxicity, or if they withdrew early because of toxicity from the platinum-doublet chemotherapy, entered the post-study treatment phase and continued same treatment until PD, unacceptable toxicity or death. Participants who withdrew due to PD or toxicity from placebo could not enter the post-study treatment phase. Upon PD (during either the primary or post-study treatment phase), participants had the option to be crossed over to open-label erlotinib 150 mg/day outside the study (Off-study phase).
- Erlotinib: Participants received 1250 mg/m^2 of gemcitabine IV infusion on Day 1 and 8, carboplatin 5x AUC or cisplatin 75 mg/m^2 IV infusion on Day 1 and oral erlotinib 150 mg/day from Day 15 to 28 every 4 weeks, continued for 6 cycles (28-day cycle) until PD, unacceptable toxicity or death in the primary study treatment phase. Participants who completed 6 cycles of treatment without PD or unacceptable toxicity, or if they withdrew early because of toxicity from the platinum-doublet chemotherapy, entered the post-study treatment phase and continued same treatment until PD, unacceptable toxicity or death. Participants who withdrew due to PD or toxicity from erlotinib could not enter the post-study treatment phase. Upon PD (during either the primary or post-study treatment phase), participants were treated at the discretion of the investigators' discretion (Off-study phase).
- Total: Total of all reporting groups
Arm/Group | Placebo | Erlotinib | Total
Number analyzed (Participants) | 225 | 226 | 451
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (11.08) | 57.2 (9.71) | 56.8 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 94 | 179
  Male | 140 | 132 | 272

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (PFS) Time
Description: Tumor response was evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0). PD was defined as at least a 20 percent (%) increase in the sum of longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions. PFS is the time (in months) between the date of randomization and the date of first documented disease progression or death from any cause, whichever comes first. Participants who had neither progressed nor died at the time of data cut-off or who were lost to follow-up were censored at the date of the last tumor assessment where non-progression was documented or last date of follow up for progression of disease, whichever was last. Participants without post baseline tumor assessments who were known to be alive were censored at the time of randomization. Analysis was performed using Kaplan-Meier method.
Time Frame: Randomization until PD or death (assessed at baseline and every 8 weeks thereafter until PD, death or end of study [up to approximately 1.5 years])
Population: FAS population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Erlotinib
Number analyzed (Participants) | 225 | 226
months | 6.0 [6.0 to 7.0] | 7.6 [7.0 to 8.0]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.46 to 0.70]

2. Secondary Outcome: Percentage of Participants Alive and Free From Disease Progression
Description: Tumor response was evaluated according to RECIST (version 1.0). PD was defined as at least a 20% increase in the sum of LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions.
Time Frame: as for outcome 1
Population: FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Erlotinib
Number analyzed (Participants) | 225 | 226
percentage of participants | 6.2 | 22.6

3. Secondary Outcome: Median PFS Time Based on Different Subgroups
Description: Tumor response was evaluated according to RECIST (version 1.0). PD was defined in outcome measure 1. PFS is the time (in months) between the date of randomization and the date of first documented disease progression or death from any cause, whichever comes first. Participants who had neither progressed nor died at the time of data cut-off or who were lost to follow-up were censored at the date of the last tumor assessment where non-progression was documented or last date of follow up for progression of disease, whichever was last. Participants without post baseline tumor assessments who were known to be alive were censored at the time of randomization. PFS among different subgroups of type of carcinoma, smoking habit, epidermal growth factor receptor (EGFR) mutation type, KRAS mutation type, EGFR immunohistochemistry (IHC) test result type, and EGFR fluorescent in situ hybridization (FISH) result type.
Time Frame: as for outcome 1
Population: FAS population. "n" is the number of participants evaluable under the specified category.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Erlotinib
Number analyzed (Participants) | 225 | 226
months
  Adenocarcinoma (n=168,174) | 6.5 [6 to 7] | 8.2 [8 to 11]
  Non-adenocarcinoma (n=57,52) | 5.8 [5 to 7] | 5.7 [3 to 7]
  Never smoked (n=107,112) | 6.6 [5 to 7] | 10.9 [9 to 14]
  Former/current smoker (n=118,114) | 5.9 [5.5 to 7.1] | 5.7 [4 to 7]
  EGFR mutation (n=48,49) | 6.9 [5 to 8] | 15.6 [13 to NA] — Estimate not available due to insufficient follow-up to allow estimation.
  EGFR wild-type (n=67,69) | 5.9 [5 to 7] | 7.1 [4 to 8]
  KRAS mutation (n=11,10) | 4.5 [1.9 to 7.2] | 6.0 [2.4 to 8.9]
  KRAS wild-type (n=101,101) | 6.8 [5.6 to 7.3] | 8.0 [7.5 to 10.8]
  EGFR IHC positive (n=36,40) | 6.0 [3.7 to 8.8] | 8.1 [7.4 to 11.0]
  EGFR IHC negative (n=25,12) | 6.7 [4.6 to 7.6] | 10.1 [7.6 to 15.6]
  EGFR FISH positive (n=20,14) | 5.9 [2.2 to 9.3] | 12.9 [9.4 to NA] — Estimate not available due to insufficient follow-up to allow estimation.
  EGFR FISH negative (n=23,25) | 6.0 [4.6 to 8.8] | 7.5 [6.2 to 9.7]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib; PFS in adenocarcinoma subgroup; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.39 to 0.64]
Statistical Analysis 2: Comparison: Placebo vs Erlotinib; PFS in non-adenocarcinoma subgroup; Test type: Superiority or Other; p = 0.579, Log Rank; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.60 to 1.33]
Statistical Analysis 3: Comparison: Placebo vs Erlotinib; PFS in never smoked subgroup; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.39, 95% CI 2-sided [0.28 to 0.53]
Statistical Analysis 4: Comparison: Placebo vs Erlotinib; PFS in former/current smoker subgroup; Test type: Superiority or Other; p = 0.2067, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.64 to 1.10]
Statistical Analysis 5: Comparison: Placebo vs Erlotinib; PFS in subgroup EGFR mutation; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.21, 95% CI 2-sided [0.12 to 0.35]
Statistical Analysis 6: Comparison: Placebo vs Erlotinib; PFS in subgroup EGFR wild-type; Test type: Superiority or Other; p = 0.7511, Log Rank; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.67 to 1.34]
Statistical Analysis 7: Comparison: Placebo vs Erlotinib; PFS in subgroup KRAS mutation; Test type: Superiority or Other; p = 0.3169, Log Rank; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.25 to 1.58]
Statistical Analysis 8: Comparison: Placebo vs Erlotinib; PFS in subgroup KRAS wild-type; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.37 to 0.70]
Statistical Analysis 9: Comparison: Placebo vs Erlotinib; PFS in subgroup EGFR IHC positive; Test type: Superiority or Other; p = 0.0091, Log Rank; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.31 to 0.86]
Statistical Analysis 10: Comparison: Placebo vs Erlotinib; PFS in subgroup EGFR IHC negative; Test type: Superiority or Other; p = 0.0179, Log Rank; Hazard Ratio (HR) = 0.40, 95% CI 2-sided [0.18 to 0.88]
Statistical Analysis 11: Comparison: Placebo vs Erlotinib; PFS in subgroup EGFR FISH positive; Test type: Superiority or Other; p = 0.0017, Log Rank; Hazard Ratio (HR) = 0.26, 95% CI 2-sided [0.11 to 0.64]
Statistical Analysis 12: Comparison: Placebo vs Erlotinib; PFS in subgroup EGFR FISH negative; Test type: Superiority or Other; p = 0.1880, Log Rank; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.37 to 1.22]

4. Secondary Outcome: Median Overall Survival (OS) Time-Overall and Among Different Subgroups
Description: OS was defined as the time between the date of randomization and the date of death from any cause. Participants for whom no death was captured on the clinical database were censored at the most recent date they were known to be alive. Participants with no post baseline information were censored at the time of randomization. OS among different subgroups of type of carcinoma, smoking habit, EGFR mutation type, KRAS mutation type, EGFR IHC test result type, and EGFR FISH result type. Analysis was performed using Kaplan-Meier method.
Time Frame: Randomization until death (assessed at baseline and every 8 weeks thereafter until death or end of study [up to approximately 5.5 years])
Population: FAS population. "n" is the number of participants evaluable under the specified category.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Erlotinib
Number analyzed (Participants) | 225 | 226
months
  Overall participants (n=225,226) | 15.2 [12.7 to 17.5] | 18.2 [16.3 to 20.8]
  Adenocarcinoma (n=168,174) | 15.8 [13.6 to 18.5] | 20.9 [18.3 to 25.9]
  Non-adenocarcinoma (n=57,52) | 12.4 [9.9 to 16.8] | 10.3 [7.6 to 13.0]
  Never smoked (n=107,112) | 17.5 [14.8 to 21.7] | 25.9 [21.6 to 32.4]
  Current/former smoker (n=118,114) | 13.0 [11.0 to 15.8] | 13.0 [10.0 to 16.3]
  EGFR mutation (n=48,49) | 20.6 [14.2 to 31.1] | 30.3 [22.2 to 37.1]
  EGFR wild-type (n=67,69) | 12.2 [8.9 to 14.7] | 14.9 [12.2 to 18.2]
  KRAS mutation (n=11,10) | 11.2 [5.7 to 16.5] | 17.5 [6.3 to 18.8]
  KRAS wild-type (n=101,101) | 14.1 [12.4 to 18.2] | 18.1 [15.4 to 22.2]
  EGFR IHC positive (n=36,40) | 15.2 [12.1 to 19.6] | 18.6 [16.3 to 32.4]
  EGFR IHC negative (n=25,12) | 12.5 [7.8 to 19.8] | 21.9 [14.3 to NA] — Estimate not available due to insufficient follow-up to allow estimation.
  EGFR FISH positive (n=20,14) | 17.7 [8.9 to 23.8] | 43.1 [18.6 to NA] — Estimate not available due to insufficient follow-up to allow estimation.
  EGFR FISH negative (n=23,25) | 12.5 [10.3 to 16.0] | 16.7 [13.1 to 22.4]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib; OS in overall participants (FAS population); Test type: Superiority or Other; p = 0.1213, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.70 to 1.04]
Statistical Analysis 2: Comparison: Placebo vs Erlotinib; OS in subgroup adenocarcinoma; Test type: Superiority or Other; p = 0.0356, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.62 to 0.98]
Statistical Analysis 3: Comparison: Placebo vs Erlotinib; OS in subgroup non-adenocarcinoma; Test type: Superiority or Other; p = 0.1157, Log Rank; Hazard Ratio (HR) = 1.37, 95% CI 2-sided [0.92 to 2.03]
Statistical Analysis 4: Comparison: Placebo vs Erlotinib; OS in subgroup never smoked; Test type: Superiority or Other; p = 0.0056, Log Rank; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.49 to 0.89]
Statistical Analysis 5: Comparison: Placebo vs Erlotinib; OS in subgroup current/former smoker; Test type: Superiority or Other; p = 0.3473, Log Rank; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.87 to 1.50]
Statistical Analysis 6: Comparison: Placebo vs Erlotinib; OS in subgroup EGFR mutation; Test type: Superiority or Other; p = 0.1614, Log Rank; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.45 to 1.14]
Statistical Analysis 7: Comparison: Placebo vs Erlotinib; OS in subgroup EGFR wild-type; Test type: Superiority or Other; p = 0.1691, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.55 to 1.11]
Statistical Analysis 8: Comparison: Placebo vs Erlotinib; OS in subgroup KRAS mutation; Test type: Superiority or Other; p = 0.1415, Log Rank; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.19 to 1.28]
Statistical Analysis 9: Comparison: Placebo vs Erlotinib; OS in subgroup KRAS wild-type; Test type: Superiority or Other; p = 0.1447, Log Rank; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.59 to 1.08]
Statistical Analysis 10: Comparison: Placebo vs Erlotinib; OS in EGFR IHC positive; Test type: Superiority or Other; p = 0.0310, Log Rank; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.35 to 0.96]
Statistical Analysis 11: Comparison: Placebo vs Erlotinib; OS in subgroup EGFR IHC negative; Test type: Superiority or Other; p = 0.0581, Log Rank; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.21 to 1.05]
Statistical Analysis 12: Comparison: Placebo vs Erlotinib; OS of subgroup EGFR FISH positive; Test type: Superiority or Other; p = 0.0063, Log Rank; Hazard Ratio (HR) = 0.32, 95% CI 2-sided [0.14 to 0.75]
Statistical Analysis 13: Comparison: Placebo vs Erlotinib; OS of subgroup EGFR FISH negative; Test type: Superiority or Other; p = 0.3268, Log Rank; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.40 to 1.36]

5. Secondary Outcome: Percentage of Participants Alive at the End of Study-Overall and Among Different Subgroups
Time Frame: as for outcome 4
Population: FAS population. "n" is the number of participants evaluable under the specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Erlotinib
Number analyzed (Participants) | 225 | 226
percentage of participants
  Overall participants (n=225,226) | 13.3 | 15.9
  Adenocarcinoma (n=168,174) | 14.9 | 19.5
  Non-adenocarcinoma (n=57,52) | 8.8 | 3.8
  Never smoked (n=107,112) | 13.1 | 23.2
  Current/former smoker (n=118,114) | 13.6 | 8.8
  EGFR mutation (n=48,49) | 22.9 | 30.6
  EGFR wild-type (n=67,69) | 7.5 | 10.1
  KRAS mutation (n=11,10) | 0.0 | 20.0
  KRAS wild-type (n=101,101) | 14.9 | 17.8
  EGFR IHC positive (n=36,40) | 11.1 | 25.0
  EGFR IHC negative (n=25,12) | 8.0 | 33.3
  EGFR FISH positive (n=20,14) | 10.0 | 42.9
  EGFR FISH negative (n=23,25) | 13.0 | 16.0

6. Secondary Outcome: Non-Progression Rate: Percentage of Participants With a Confirmed Best Overall Response of Either Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) for At Least 16 Weeks
Description: Tumor response was evaluated according to RECIST (version 1.0). CR is defined as the disappearance of all target and non-target lesions and normalization of tumor marker level; PR is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the screening sum LD; SD for target lesions is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started and SD for non-target lesions defined as persistence of 1 or more non-target lesion(s) or/and maintenance of tumor marker level above the normal limits. Responses were confirmed with repeated assessment 4 weeks after initial response was observed.
Time Frame: as for outcome 1
Population: FAS population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Erlotinib
Number analyzed (Participants) | 225 | 226
percentage of participants | 64.4 [57.8 to 70.7] | 67.3 [60.7 to 73.3]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib; Difference in non-progression response rates; Test type: Superiority or Other; p = 0.5289, Chi-squared; Mean Difference (Final Values) = 2.81, 95% CI 2-sided [-6.2 to 11.8]

7. Secondary Outcome: Objective Response Rate: Percentage of Participants With a Confirmed Best Overall Response of CR or PR
Description: Tumor response was evaluated according to RECIST (version 1.0). CR is defined as the disappearance of all target and non-target lesions and normalization of tumor marker level; PR is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the screening sum LD. Responses were confirmed with repeated assessment 4 weeks after initial response was observed.
Time Frame: as for outcome 1
Population: FAS population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Erlotinib
Number analyzed (Participants) | 225 | 226
percentage of participants | 17.8 [13.0 to 23.4] | 42.9 [36.4 to 49.7]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib; Difference in objective response rates; Test type: Superiority or Other; p < 0.0001, Chi-squared; Mean Difference (Final Values) = 25.14, 95% CI 2-sided [16.7 to 33.5]

8. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time between the date of first documented response (CR or PR, as determined by the RECIST criteria) and the date of first documented PD or death. Participants who did not progress or die after they had a confirmed response (CR or PR) were censored at the date of their last tumor assessment where non-progression was documented or last date of follow-up for progression of disease, whichever was last. CR and PR are defined in Outcome Measure 7.
Time Frame: as for outcome 1
Population: FAS population participants who were responders (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Erlotinib
Number analyzed (Participants) | 40 | 97
months | 5.6 [5 to 6] | 10.3 [7 to 13]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.32, 95% CI 2-sided [0.21 to 0.50]

9. Secondary Outcome: Time to Progression
Description: Time to progression is defined as the time between the date of randomization and the date of the first documented disease progression. Participants who have not progressed at the time of study completion (or data cut off) or who were lost to follow up were censored at the date of the last tumor assessment where non-progression was documented or last date of follow-up for progression of disease, whichever was latest. PD was defined as at least a 20% increase in the sum of LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions. Participants with no post baseline tumor assessments were censored at the time of randomization. Analysis was performed using Kaplan-Meier method.
Time Frame: Randomization until PD (assessed at baseline and every 8 weeks thereafter until PD or end of study [up to approximately 1.5 years])
Population: FAS population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Erlotinib
Number analyzed (Participants) | 225 | 226
months | 6.5 [6 to 7] | 7.9 [7 to 9]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.45 to 0.69]

10. Secondary Outcome: Percentage of Participants With Symptomatic Progression Assessed Using the Lung Cancer Subscale (LCS)
Description: LCS scores were obtained from a 7-item questionnaire from the Functional Assessment of Cancer Therapy - Lung (FACT-L) (version 4.0). Participants responded to questions such as shortness of breath, cough, tightness in chest, breathing difficulty, appetite loss, weight loss and unclear thinking; on a 5-point scale from 0-4, where 0 equaled (=) "not at all" and 4 = "very much." The participants' responses were summed to result in an overall score, scores range on a scale of 0 (most symptomatic) to 28 (asymptomatic); higher score indicates fewer symptoms. A clinically meaningful decline used to determine symptomatic progression in this study was at least a three point decline in LCS score from baseline. Participants without symptomatic progression at the time of analysis were censored at the time of the last FACT-L assessment.
Time Frame: Baseline, Day 1 of Cycles 3 and 5, Day 1 of post-study Visits 1 and 2 until end of study medication administration or PD (up to approximately 1.5 years)
Population: FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Erlotinib
Number analyzed (Participants) | 225 | 226
percentage of participants | 72.4 | 66.4

11. Secondary Outcome: Time to Symptomatic Progression
Description: Time to symptomatic progression was the time from randomization until the earlier of a clinically meaningful decline from baseline in LCS score, or death on study. LCS scores were obtained from a 7-item questionnaire from the FACT-L (version 4.0). Participants responded to questions such as shortness of breath, cough, tightness in chest, breathing difficulty, appetite loss, weight loss and unclear thinking; on a 5-point scale from 0-4, where 0 = "not at all" and 4 = "very much." The participants' responses were summed to result in an overall score, scores range on a scale of 0 (most symptomatic) to 28 (asymptomatic); higher score indicates fewer symptoms. A clinically meaningful decline used to determine symptomatic progression in this study was at least a three point decline in LCS score from baseline. Participants without symptomatic progression at the time of analysis were censored at the time of the last FACT-L assessment. Analysis was performed using Kaplan-Meier method.
Time Frame: as for outcome 10
Population: FAS population.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Placebo | Erlotinib
Number analyzed (Participants) | 225 | 226
months | 6.6 [6 to 9] | 7.2 [6 to 10]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib; Test type: Superiority or Other; p = 0.0364, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.63 to 0.99]

12. Secondary Outcome: Percentage of Participants With Deterioration in Trial Outcome Index (TOI) Using FACT-L Version 4.0
Description: TOI was defined as the sum of the scores of the Physical Well-Being (PWB), Functional Well-Being (FWB), and LCS. PWB, FWB, and LCS scores were obtained from 7-item questionnaires from the FACT-L (Version 4.0). Participants responded to questions on a 5-point scale from 0-4, where 0 = "not at all" and 4 = "very much." The participants' responses were summed to result in an overall score, scores range on a scale of 0 to 84; higher score indicates better physical aspects of quality of life (QoL). A clinically meaningful decline used to determine deterioration in TOI was greater than or equal to (≥) 6-point decline from baseline. Participants without deterioration in TOI at the time of analysis were censored at the time of the last FACT-L assessment.
Time Frame: as for outcome 10
Population: FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Erlotinib
Number analyzed (Participants) | 225 | 226
percentage of participants | 75.6 | 65.9

13. Secondary Outcome: Time to Deterioration in TOI Using FACT-L Version 4.0
Description: Time to deterioration in TOI is defined as time from randomization until the earlier of a clinically meaningful decline from baseline in TOI or death on study. TOI is defined as the sum of the scores of the PWB, FWB, and LCS. PWB, FWB, and LCS scores were obtained from 7-item questionnaires from the FACT-L (Version 4.0). Participants responded to questions on a 5-point scale from 0-4, where 0 = "not at all" and 4 = "very much." The participants' responses were summed to result in an overall score, scores range on a scale of 0 to 84; higher score indicates better physical aspects of QoL. A clinically meaningful decline used to determine deterioration in TOI was ≥6-point decline from baseline. Participants without deterioration in TOI at the time of analysis were censored at the time of the last FACT-L assessment. Analysis was performed using Kaplan-Meier method.
Time Frame: as for outcome 10
Population: FAS population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Erlotinib
Number analyzed (Participants) | 225 | 226
months | 5.6 [4 to 7] | 6.3 [5 to 8]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib; Test type: Superiority or Other; p = 0.0181, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.61 to 0.96]

14. Secondary Outcome: Percentage of Participants With Deterioration in Quality of Life (QOL) Using FACT-L Version 4.0
Description: Total FACT-L score was defined as the sum of the TOI, Social Well Being (SWB) and EWB of the FACT-L questionnaires. TOI (PWB + FWB + LCS), SWB and EWB scores were obtained from 7-item (6-item in the case of EWB) questionnaires from the FACT-L (Version 4.0). Participants responded to questions on a 5-point scale from 0-4, where 0 = "not at all" and 4 = "very much." The participants' responses were summed to result in an overall score, scores range on a scale of 0 to 136; higher score indicates better QoL. A clinically meaningful decline used to determine deterioration in QoL was ≥6-point decline from baseline. Participants without deterioration in QoL at the time of analysis were censored at the time of the last FACT-L assessment.
Time Frame: as for outcome 10
Population: FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Erlotinib
Number analyzed (Participants) | 225 | 226
percentage of participants | 79.6 | 70.4

15. Secondary Outcome: Time to Deterioration in QOL Using FACT-L Version 4.0
Description: Time to deterioration in QoL is defined as time from randomization until the earlier of a clinically meaningful decline from baseline in Total FACT-L or death on study. Total FACT-L score was defined as the sum of the TOI, SWB and EWB of the FACT-L questionnaires. TOI (PWB + FWB + LCS), SWB and EWB scores were obtained from 7-item (6-item in the case of EWB) questionnaires from the FACT-L (Version 4.0). Participants responded to questions on a 5-point scale from 0-4, where 0 = "not at all" and 4 = "very much." The participants' responses were summed to result in an overall score, scores range on a scale of 0 to 136; higher score indicates better QoL. A clinically meaningful decline used to determine deterioration in QoL was ≥6-point decline from baseline. Participants without deterioration in QoL at the time of analysis were censored at the time of the last FACT-L assessment. Analysis was performed using Kaplan-Meier method.
Time Frame: as for outcome 10
Population: FAS population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Erlotinib
Number analyzed (Participants) | 225 | 226
months | 4.5 [4 to 6] | 5.6 [4 to 7]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib; Test type: Superiority or Other; p = 0.0035, Log Rank; Hazard Ratio, log = 0.73, 95% CI 2-sided [0.59 to 0.90]

16. Secondary Outcome: Median Follow-up Time During the Study
Description: Median follow-up was calculated using 'Reverse Kaplan-Meier' analysis for Overall survival.
Time Frame: Randomization until PD or death (assessed at baseline and every 8 weeks thereafter until PD, death or end of study [up to approximately 5.5 years])
Population: FAS population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Erlotinib
Number analyzed (Participants) | 225 | 226
months | 50.3 [47.6 to 52.5] | 50.2 [48.2 to 51.7]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib; Test type: Superiority or Other; p = 0.9130, Log Rank; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.60 to 1.59]

ADVERSE EVENTS:
Time Frame: Up to 28 days after the last dose in the primary and post study treatment phases of the study (up to approximately 5.5 years)
Arm/Group | Placebo | Erlotinib
Serious Adverse Events (participants affected / at risk) | 76/222 | 70/226
Other Adverse Events (participants affected / at risk) | 217/222 | 223/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=222) | Erlotinib (N=226)
Anaemia (Blood and lymphatic system disorders) | 26 | 22
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 10
Neutropenia (Blood and lymphatic system disorders) | 2 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2
Bone marrow failure (Blood and lymphatic system disorders) | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Pneumonia (Infections and infestations) | 9 | 7
Cellulitis (Infections and infestations) | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 2
Pneumonia bacterial (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 1 | 2
Appendicitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Pneumonia viral (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 0 | 1
Gastroenteritis bacterial (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Oesophageal compression (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 3
Asthenia (General disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Thrombosis in device (General disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Paraparesis (Nervous system disorders) | 0 | 1
Pyramidal tract syndrome (Nervous system disorders) | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 2
White blood cell count decreased (Investigations) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal ischaemia (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 3
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Transient psychosis (Psychiatric disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Superior vena cava occlusion (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=222) | Erlotinib (N=226)
Neutropenia (Blood and lymphatic system disorders) | 110 | 114
Leukopenia (Blood and lymphatic system disorders) | 51 | 42
Anaemia (Blood and lymphatic system disorders) | 96 | 87
Thrombocytopenia (Blood and lymphatic system disorders) | 46 | 45
Nausea (Gastrointestinal disorders) | 92 | 90
Vomiting (Gastrointestinal disorders) | 68 | 69
Diarrhoea (Gastrointestinal disorders) | 34 | 69
Constipation (Gastrointestinal disorders) | 46 | 47
Stomatitis (Gastrointestinal disorders) | 8 | 27
Mouth ulceration (Gastrointestinal disorders) | 2 | 15
Dyspepsia (Gastrointestinal disorders) | 14 | 4
Abdominal distension (Gastrointestinal disorders) | 5 | 13
Rash (Skin and subcutaneous tissue disorders) | 72 | 142
Alopecia (Skin and subcutaneous tissue disorders) | 51 | 41
Pruritus (Skin and subcutaneous tissue disorders) | 21 | 27
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 12 | 33
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 34
Fatigue (General disorders) | 60 | 55
Pyrexia (General disorders) | 25 | 37
Asthenia (General disorders) | 16 | 16
Mucosal inflammation (General disorders) | 13 | 24
Chest pain (General disorders) | 21 | 24
Malaise (General disorders) | 10 | 12
Decreased appetite (Metabolism and nutrition disorders) | 92 | 79
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 35 | 37
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 25
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 19 | 18
Hiccups (Respiratory, thoracic and mediastinal disorders) | 14 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 13
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 13
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 12
Alanine aminotransferase increased (Investigations) | 19 | 16
White blood cell count decreased (Investigations) | 13 | 10
Aspartate aminotransferase increased (Investigations) | 12 | 11
Weight decreased (Investigations) | 7 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 22
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 8
Dizziness (Nervous system disorders) | 20 | 23
Headache (Nervous system disorders) | 18 | 14
Insomnia (Psychiatric disorders) | 37 | 46
Upper respiratory tract infection (Infections and infestations) | 9 | 16
Nasopharyngitis (Infections and infestations) | 12 | 10
Paronychia (Infections and infestations) | 0 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.